CLINICAL TRIAL: NCT01080014
Title: The Multiple Sclerosis Functional Composite (MSFC) in the Follow-up of MS Patients: Correlation With the Expanded Disability Status Scale (EDSS) Among Different Clinical Forms in Argentina
Brief Title: Correlation Between Multiple Sclerosis Functional Composite (MSFC) and Expanded Disability Status Scale (EDSS) in Patients With Multiple Sclerosis (MS) in Argentina
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200077_502
Record Dates: First submitted 2010-02-24; First posted 2010-03-03 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing-remitting multiple sclerosis (RRMS); primary progressive multiple sclerosis (PPMS); secondary progressive multiple sclerosis (SPMS); Multiple Sclerosis Functional Composite (MSFC); Expanded Disability Status Scale (EDSS)
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This observational study is being conducted to evaluate the usefulness of the MSFC and its relationship with EDSS scores in subjects with MS in Argentina.

DETAILED DESCRIPTION:
This observational, open-label study is being conducted to correlate change in EDSS score with the change in MSFC scores at the end of a 2-year follow-up period for subjects with MS in Argentina. Measurement of disability is an indispensable parameter in assessing the efficacy of experimental therapeutic agents in MS as well as in trying to determine possible individual evolution of the disease. Clinical scales are being used as primary or secondary outcome measures for recording disease progression in clinical trials. Kurtzke's EDSS is still used as a gold standard for measuring impairment and disability in MS. The MSFC is an examination-based quantitative scoring of neurological impairment. This study aims to establish a correlation between the usefulness of both scales.

OBJECTIVES

Primary Objective:

* To evaluate the change in MSFC score with change in EDSS scores at end of 2 year follow-up period for subjects with MS in Argentina

Secondary Objectives:

* To evaluate the cross-sectional correlations in MSFC score at baseline and at 24 months with EDSS score at baseline and at 24 months
* To describe the MSFC score for MS phenotype in this population
* To evaluate the predictive validity of MSFC score of a subsequent EDSS change in a subgroup of MS patients in Argentina

ELIGIBILITY:
Inclusion Criteria:

* Subjects with definite diagnosis of MS, according to McDonald's criteria
* All clinical types: relapsing-remitting MS (RRMS), primary progressive MS (PPMS) and secondary progressive MS (SPMS). Stable disease course without any relapse for at least the previous 3 months
* Subjects treated or not with disease modifying drugs
* Ages between 18 and 65 years and is capable of understanding and complying with protocol requirements
* Subject has a stable residence with no planned move during the entire investigation period

Exclusion Criteria:

* Life expectancy less than 5 years at admission
* Diagnosis of clinically isolated syndrome (CIS)
* Other clinical conditions that mimic MS
* Psychiatric diseases
* Alcohol or drug abuse
* Pregnancy
* The subject is unwilling or unable to comply with the protocol or scheduled appointments
* Subject is unable to understand the language in which the approved informed consent is written
* The subject is a study site employee, or an immediate family member (i.e., spouse, parent, child, sibling) of a study site employee, involved in conduct of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with MS in 20 sites across Argentina
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2008-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
- Evaluation of correlations between changes over time | Baseline and two years
  - Evaluation of correlations between changes over time for MSFC composite score and arm, leg and cognitive MSFC scores versus EDSS score changes over the same periods

SECONDARY OUTCOMES:
To evaluate the predictive validity of MSFC score of a subsequent EDSS change in a subgroup of MS patients | Baseline, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Roberto Rosa, PhD, Principal Investigator — PhD Neurologist, Unaffiliated
Locations (1):
- Dr. Roberto Rosa, Buenos Aires, Argentina